CLINICAL TRIAL: NCT02613624
Title: Formative Research to Develop an Intervention Package for Promotion of Kangaroo Mother Care for Low Birth Weight and Preterm Infants in a Community: In Preparation for a Randomized Controlled Trial to Examine Impact of Community Kangaroo Mother Care on Neonatal and Early Infant Mortality
Brief Title: Formative Research to Develop an Intervention Package to Promote Practice of Kangaroo Mother Care for Low Birth Weight and Preterm Infants in a Community (CKMC)
Acronym: CKMC
Status: Completed | Type: Observational
Sponsor: Society for Applied Studies (Other)
Collaborators: Centre For International Health (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/1913/REK vest
Record Dates: First submitted 2015-10-12; First posted 2015-11-24 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Low-Birth-Weight
Keywords: KMC in community

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is being conducted to develop an intervention to assess the feasibility of implementing Kangaroo Mother Care (KMC) for low birth weight (LBW) and preterm babies in a community setting. A prototype intervention package will be developed using information obtained from in-depth interviews, focus group discussions and other qualitative research techniques. These interviews will help us identify current behaviours, barriers to adoption of KMC and effective ways to promote KMC in the community. The prototype intervention will be refined by conducting acceptability studies (household trials) with few mothers. The study team are identifying LBW and preterm infants, demonstrating to mothers how to practice KMC and following up till KMC is stopped. The process is being documented using observations and interviews. Information is obtained on acceptability of KMC, number of hours per day and number of days KMC was given, breastfeeding practices and support provided by other family members.

ELIGIBILITY:
Inclusion Criteria:

* Low birth weight or preterm newborns

Exclusion Criteria:

* Babies with hospitalization criteria
* unable to feed or weight less than 1500 grams at birth

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Rural and semi urban population of two primary health centre areas in two districts of the state of Haryana, India.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of community based KMC | 1 year
  To determine whether community KMC is feasible to implement in the study setting and if so, can high enough adoption rates be achieved. This will be ascertained by documenting proportion of mothers doing KMC, number of hours each day and number of days skin to skin contact is given.
Define intervention package | 1 year
  To define an intervention package, including the most effective way(s) to promote KMC in the study setting.

SECONDARY OUTCOMES:
Perceptions and practices of maternal and newborn care | 1 year
  To ascertain perceptions, beliefs and practices around pregnancy, delivery and maternal and newborn care. Qualitative research methods such as focus group discussions, in-depth interviews and observations using open ended questionnaires, interview guides and checklists will be used.
Social norms around birthing practices | 1 year
  To identify social norms around birthing practices for normal, LBW infants and preterms. Qualitative research methods such as focus group discussions, in-depth interviews and observations using open ended questionnaires, interview guides and checklists will be used.
Awareness and perception around KMC | 1 year
  To ascertain awareness and perceptions around KMC. Qualitative research methods such as focus group discussions, in-depth interviews and observations using open ended questionnaires, interview guides and checklists will be used.
Promotion of KMC | 1 year
  To identify ways to promote KMC in the community.

CONTACTS AND LOCATIONS:
Overall Officials: Sarmila Mazumder, MBBS, PhD, Principal Investigator — Centre for Health Research and Development, Society for Applied Studies, New Delhi
Locations (1):
- CHRD, Society for Applied Studies, Palwal, Haryana, India